CLINICAL TRIAL: NCT04845516
Title: Efficacy and Tolerance of Therapeutic Apheresis in Paediatric Neurology: a Retrospective French Multicenter Study
Brief Title: Efficacy and Tolerance of Therapeutic Apheresis in Paediatric Neurology: a French Multicenter Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0084
Record Dates: First submitted 2021-02-16; First posted 2021-04-15 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Apheresis Related Complication
Keywords: Children; therapeutic exchange; neuropediatric; immunoadsorption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- plasma exchange: All patients underwent plasma exchanges between 2014 and 2019 for a neuropediatric pathology
  Interventions: Other: Efficacy of apheresis
- immunoadsorption: All patients who underwent immunoadsorptions between 2014 and 2019 for a neuropediatric pathology
  Interventions: Other: Efficacy of apheresis

INTERVENTIONS:
Other: Efficacy of apheresis — Efficacy of apheresis

SUMMARY:
After developing in pediatric hematology and nephrology, therapeutic apheresis is increasingly used in pediatric neurology despite a sparse level of evidence.

There are a few retrospective series with a small number of patients, concerning mainly autoimmune diseases (encephalitis, myasthenia gravis, polyradiculoneuritis).

The objective of this work is to study therapeutic apheresis (including plasma exchange and immunoadsorption) among french neuropediatric tertiary centers and to prove that this treatment modality is effective and well tolerated in pediatric neurology diseases.

DETAILED DESCRIPTION:
Multicenter medical data collection :

* Montpellier
* Toulouse
* Bordeaux
* Marseille
* Nancy
* Paris Kremlin Bicêtre
* Paris Robert Debré
* Paris Necker
* Paris Trousseau
* Lyon
* Besançon
* Rennes
* Reims
* Strasbourg
* La Réunion
* Nantes
* Tours

ELIGIBILITY:
Inclusion criteria:

* Children under 18.
* Supported in a participating CHU between 2014 and 2019.
* Having benefited from therapeutic apheresis (plasma exchanges and immunoadsorption) in a neuropediatric indication

Exclusion criteria:

- Family or patient refusal to participate

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18, Supported in a participating CHU between 2014 and 2019 and Having benefited from therapeutic apheresis (plasma exchanges and immunoadsorption) in a neuropediatric indication
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
global neurological efficacy of therapeutic apheresis as assessed | through study completion, an average of 2 years
  lobal neurological efficacy of therapeutic apheresis as assessed by modified rankin score Modifed Rankin score, ranging from 0 (no symptoms) to 6 (death)

SECONDARY OUTCOMES:
Incidence of therapeutic apheresis adverse events as assessed | through study completion, an average of 2 years
  tIncidence of therapeutic apheresis adverse events as assessed by low blood tension rate, transfusion rate, infection rate, hypocalcaemia rate, thrombosis rate, allergy rate, anemia rate, hemostasis disorders rate).
Incidence of adjuvant treatments | through study completion, an average of 2 years
  Incidence of adjuvant treatments (corticosteroid therapy, immunoglobulins, immunosuppressants),
Incidence of hospitalization in intensive care | through study completion, an average of 2 years
  Incidence of hospitalization in intensive care, intubation rate
Description of the therapeutic apharesis modalities | through study completion, an average of 2 years
  number of procedures
Description of the therapeutic apharesis modalities | through study completion, an average of 2 years
  exchanged volume (in plasma volume percentage) for each procedure
Description of the therapeutic apharesis modalities | through study completion, an average of 2 years
  type of separation et number of participants with ttt-related advesre events
Description of the therapeutic apharesis modalities | through study completion, an average of 2 years
  type of replacement solution (isotonic saline, albumin, fresh frozen plasma)
Number of participitants with treatment-related adverse events | during procedures
  rate of arterial hypotension (< age standards and and requiring isotonic saline bolus, for each patient and for procedure)
Number of participitants with treatment-related adverse events | during procedures
  rate of hypocalcemia (ionized calcium <1,1 mmol/L, for each patient and for each procedure)
Number of participitants with treatment-related adverse events | during procedures
  rate of hypoalbuminemiafor for each patient and for each procedure)
Number of participitants with treatment-related adverse events | during procedures
  rate of thrombosis (confirmed by a CT scan or ultrasound, for each patient)
Number of participitants with treatment-related adverse events | during procedures
  rate of infections related catheter (for each patient)
Number of participitants with treatment-related adverse events | during procedures
  rate of allergics reactions (for each patient and for each procedure)
Number of participitants with treatment-related adverse events | during procedures
  rate of anemia (Hb < 7,0 g/dL, for each patient)
Number of participitants with treatment-related adverse events | during procedures
  rate of transfusion (for each patient)
Number of participitants with treatment-related adverse events | during procedures
  rate of haemostasis disorder (platelets < 100 <G/L ; TQ < 40 % ; fibrinogen < 1 G/L ; (for each patient and for each procedure)
Number of participitants with treatment-related adverse events | during procedures
  rate of death

CONTACTS AND LOCATIONS:
Overall Officials: Maxime colmard, résident, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC